CLINICAL TRIAL: NCT01293149
Title: The Effects of Clonidine on Postoperative Analgesia After Single Shot Femoral Nerve Block Following Arthroscopic Knee Surgery in Children
Brief Title: Clonidine in Femoral Nerve Block Surgery in Children
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Amod Sawardekar, MD/ Clinical Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB11-00075
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Other Reconstructive Surgery
Keywords: knee, reconstructive surgery; femoral nerve block
MeSH Terms: interventions — Ropivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine plus clonidine (Experimental): Ropivacaine plus clonidine for femoral block
  Interventions: Drug: Clonidine
- Ropivacaine (Active Comparator): Ropivacaine alone for femoral block
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — ropivacaine 0.2% 0.5 ml/kg (max 20 ml)
  Arms: Ropivacaine
Drug: Clonidine — clonidine 1 mcg/kg AND ropivacaine 0.2% 0.5 ml/kg (max 20 ml)
  Arms: Ropivacaine plus clonidine

SUMMARY:
Knee arthroscopy is a common surgical procedure in pediatrics in which the knee joint is visualized through a small camera to help diagnose and treat knee problems. This procedure is commonly accomplished with the use of general anesthesia. Regional anesthesia is commonly completed with a single injection of local anesthetic around the femoral nerve to provide pain relief for several hours following knee arthroscopy. The intent of this study is to examine the effects of clonidine in addition to local anesthetics for femoral nerve blockade in providing children and adolescents post-operative analgesia. The investigators hypothesize the addition of low dose clonidine (1 mcg/kg) provides an additional 4 hours of post operative analgesia following arthroscopic knee surgery and reduces post-operative opiate requirement.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) functional status I or II
* Patients scheduled for arthroscopic knee surgery only

Exclusion Criteria:

* Patients with history of chronic opioid therapy, central or peripheral neuropathy, contraindications to regional anesthesia, history of allergy to clonidine or ropivicaine, or anterior cruciate ligament reconstructive surgery in addition to knee arthroscopy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  The primary end-point of the study is time from performance of femoral nerve block to onset of pain in the distribution of the femoral nerve.

SECONDARY OUTCOMES:
Heart rate | 15, 30 & 60 mins. post-op
Blood pressure | 15, 30 & 60 mins. post-op
Oxygen saturation | 15, 30 & 60 mins. post-op

CONTACTS AND LOCATIONS:
Overall Officials: Amod Sawardekar, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States